CLINICAL TRIAL: NCT03422653
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of Intravenous CR845 in Hemodialysis Patients With Moderate-to-Severe Pruritus, With a 52-Week Open Label Extension
Brief Title: A Study to Evaluate the Safety and Efficacy of CR845 in Hemodialysis Patients With Moderate-to-Severe Pruritus (KALM-1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845-CLIN3102
Record Dates: First submitted 2018-01-25; First posted 2018-02-06 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-03

CONDITIONS: Uremic Pruritus
Keywords: CR845; Pruritus; Chronic Itch; Itch; Itching; difelikefalin; Hemodialysis; Uremic Pruritus; Dialysis; CKD; CKD-associated pruritus; CKD-aP; ESRD (end stage renal disease); KALM; Chronic Kidney Disease; Kidney failure, chronic; Kidney dysfunction; Generalized pruritus
MeSH Terms: conditions — Pruritus; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — difelikefalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CR845 0.5mcg/kg (Active Comparator): IV CR845 0.5 mcg/kg administered after each dialysis session (3 times/week)
  Interventions: Drug: CR845 0.5 mcg/kg
- Placebo (Placebo Comparator): IV Placebo administered after each dialysis session (3 times/week)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CR845 0.5 mcg/kg — IV medication delivered three times/week
  Other Names: CR845; Difelikefalin
  Arms: CR845 0.5mcg/kg
Drug: Placebo — IV medication delivered three times/week
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of intravenous (IV) CR845 at a dose of 0.5 mcg/kg administered after each dialysis session. The study includes a 12-week Double-blind Phase and a 52-week Open-label Extension Phase.

DETAILED DESCRIPTION:
Double-blind Phase The Double-blind Phase of the study will consist of a Screening Visit, a 7-day Run-in Period, a 12 week Double-blind Treatment Period, and a 2-week Discontinuation Period. Informed consent will be obtained prior to performing any study-specific procedures. The Screening Visit will occur within 7 to 28 days prior to randomization to assess eligibility.

Open-label Extension Phase Patients who received at least 30 doses of study drug (either active or placebo) during the 12-week Double-blind Treatment Period and continue to meet other eligibility criteria will have the option to receive open label CR845 for an additional 52 weeks. The Open-label Extension Phase will be comprised of the Open-label Treatment Period and the Follow-up Period.

The last dose of open-label study drug will be administered at the last dialysis visit on Week 52, or Early Termination. A final safety Follow up Visit will be conducted 7-10 days after the End of Treatment/Early Termination Visit.

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible for inclusion into the Double-blind Phase of the study, a patient must meet the following criteria:

* Has end-stage renal disease (ESRD) and has been on hemodialysis 3 times per week for at least 3 months prior to the start of screening;
* Has at least 2 single-pool Kt/V measurements ≥1.2, or at least 2 urea reduction ratio measurements ≥65%, or 1 single pool Kt/V measurement ≥1.2 and 1 urea reduction ratio measurement ≥65% on different dialysis days during the 3 months period prior to screening;
* Prior to randomization:

  * Has completed Worst Itching Intensity NRS worksheets up to 8 days prior to 1st dose;
  * Has a mean baseline Worst Itching Intensity NRS indicative of moderate to severe uremic pruritus.
* To be eligible for inclusion into the Open-label Extension Phase of the study, each patient will have to fulfill the additional key following criteria at the time of entry into the Open-label Extension Phase:

  * Has received at least 30 doses of the planned 36 doses of study drug during the Double-blind Phase of this study;
  * Continues to meet inclusion criteria.

Key Exclusion Criteria:

A patient will be excluded from the Double-blind Phase of the study if any of the following criteria are met:

* Known noncompliance with dialysis treatment that in the opinion of the investigator would impede completion or validity of the study;
* Scheduled to receive a kidney transplant during the study;
* New or change of treatment received for itch including antihistamines and corticosteroids (oral, IV, or topical) within 14 days prior to screening;
* Received another investigational drug within 30 days prior to the start of screening or is planning to participate in another clinical study while enrolled in this study;
* Has pruritus only during the dialysis session (by patient report);
* Is receiving ongoing ultraviolet B and anticipates receiving such treatment during the study;
* Participated in a previous clinical study with CR845.
* A patient will be excluded from the Open-label Extension Phase of the study if any of the additional key following criteria are met at the time of entry into the Open-label Extension Phase:

  * Completed the Double-blind Phase of this study but exhibited adverse events during the course of the Treatment Period that may preclude continued exposure to the study drug;
  * Was noncompliant with protocol procedures during the Double-blind Phase of this study which is indicative of an inability to follow protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-04-06 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Menzaghi, PhD, Study Director — Cara Therapeutics
Locations (56):
- United States (56):
  - Cara Therapeutics Study Site, Homewood, Alabama
  - Cara Therapeutics Study Site, Huntsville, Alabama
  - Cara Therapeutics Study Site, Bakersfield, California
  - Cara Therapeutics Study Site 2, Beverly Hills, California
  - Cara Therapeutics Study Site, Beverly Hills, California
  - Cara Therapeutics Study Site, Chula Vista, California
  - Cara Therapeutics Study Site, Corona, California
  - Cara Therapeutics Study Site, Escondido, California
  - Cara Therapeutics Study Site, Fountain Valley, California
  - Cara Therapeutics, La Mesa, California
  - Cara Therapeutics Study Site, Long Beach, California
  - Cara Therapeutics Study Site, Ontario, California
  - Cara Therapeutics Study Site, Riverside, California
  - Cara Therapeutics Study Site, Roseville, California
  - Cara Therapeutics Study Site, San Diego, California
  - Cara Therapeutics Study Site, San Dimas, California
  - Cara Therapeutics Study Site, Tarzana, California
  - Cara Therapeutics Study Site, Denver, Colorado
  - Cara Therapeutics Study Site, Bridgeport, Connecticut
  - Cara Therapeutics Study Site, Hartford, Connecticut
  - Cara Therapeutics Study Site, Middlebury, Connecticut
  - Cara Therapeutics Study Site 1, Coral Springs, Florida
  - Cara Therapeutics Study Site, Hialeah, Florida
  - Cara Therapeutics Study Site, Miami, Florida
  - Cara Therapeutics Study Site, Miami Gardens, Florida
  - Cara Therapeutics Study Site, Tampa, Florida
  - Cara Therapeutics Study Site, Kalamazoo, Michigan
  - Cara Therapeutics Study Site, Roseville, Michigan
  - Cara Therapeutics Study Site, Minneapolis, Minnesota
  - Cara Therapeutics Study Site, Brookhaven, Mississippi
  - Cara Therapeutics Study Site, McComb, Mississippi
  - Cara Therapeutics Study Site, Tupelo, Mississippi
  - Cara Therapeutics Study Site, Kansas City, Missouri
  - Cara Therapeutics Study Site, Las Vegas, Nevada
  - Cara Therapeutics Study Site, Eatontown, New Jersey
  - Cara Therapeutics Study Site, Albuquerque, New Mexico
  - Cara Therapeutics Study Site, Gallup, New Mexico
  - Cara Therapeutics Study Site, Fresh Meadows, New York
  - Cara Therapeutics Study Site, Great Neck, New York
  - Cara Therapeutics Study Site, The Bronx, New York
  - Cara Therapeutics Study Site, Durham, North Carolina
  - Cara Therapeutics Study Site, Canton, Ohio
  - Cara Therapeutics Study Site, Roseburg, Oregon
  - Cara Therapeutics Study Site, Chattanooga, Tennessee
  - Cara Therapeutics Study Site, Dallas, Texas
  - Cara Therapeutics Study Site, Duncanville, Texas
  - Cara Therapeutics Study Site, Greenville, Texas
  - Cara Therapeutics Study Site, Houston, Texas
  - Cara Therapeutics Study Site, Lewisville, Texas
  - Cara Therapeutics Study Site, McAllen, Texas
  - Cara Therapeutics Study Site, Mesquite, Texas
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site, Waxahachie, Texas
  - Cara Therapeutics Study Site, Chesapeake, Virginia
  - Cara Therapeutics Study Site, Hampton, Virginia
  - Cara Therapeutics Study Site, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fishbane SN, Block GA, Evenepoel P, Budden J, Morin I, Menzaghi F, Wen W, Lerma EV. Pruritus Severity and Serum Phosphate in CKD: A Post Hoc Analysis of Difelikefalin Studies. Kidney360. 2024 Sep 1;5(9):1270-1280. doi: 10.34067/KID.0000000000000520. Epub 2024 Jul 22. PMID 39037824
- [Derived] Weiner DE, Schaufler T, McCafferty K, Kalantar-Zadeh K, Germain M, Ruessmann D, Morin I, Menzaghi F, Wen W, Stander S. Difelikefalin improves itch-related sleep disruption in patients undergoing haemodialysis. Nephrol Dial Transplant. 2024 Jun 28;39(7):1125-1137. doi: 10.1093/ndt/gfad245. PMID 37968132
- [Derived] Fishbane S, Wen W, Munera C, Lin R, Bagal S, McCafferty K, Menzaghi F, Goncalves J. Safety and Tolerability of Difelikefalin for the Treatment of Moderate to Severe Pruritus in Hemodialysis Patients: Pooled Analysis From the Phase 3 Clinical Trial Program. Kidney Med. 2022 Jun 28;4(8):100513. doi: 10.1016/j.xkme.2022.100513. eCollection 2022 Aug. PMID 36039153
- [Derived] Topf J, Wooldridge T, McCafferty K, Schomig M, Csiky B, Zwiech R, Wen W, Bhaduri S, Munera C, Lin R, Jebara A, Cirulli J, Menzaghi F. Efficacy of Difelikefalin for the Treatment of Moderate to Severe Pruritus in Hemodialysis Patients: Pooled Analysis of KALM-1 and KALM-2 Phase 3 Studies. Kidney Med. 2022 Jun 28;4(8):100512. doi: 10.1016/j.xkme.2022.100512. eCollection 2022 Aug. PMID 36016762
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264
- [Derived] Fishbane S, Jamal A, Munera C, Wen W, Menzaghi F; KALM-1 Trial Investigators. A Phase 3 Trial of Difelikefalin in Hemodialysis Patients with Pruritus. N Engl J Med. 2020 Jan 16;382(3):222-232. doi: 10.1056/NEJMoa1912770. Epub 2019 Nov 8. PMID 31702883

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study includes a Double-blind Phase, an Open-label Extension Phase, and a Follow-up Period. Patients who received at least 30 doses of study drug (either active or placebo) during the 12-week Double-blind Treatment Period and continue to meet other eligibility criteria will be eligible to receive open-label CR845 for an additional 52 weeks.
Groups:
- Double-blind CR845 0.5mcg/kg; Open-label CR845 0.5 mcg/kg: IV CR845 0.5 mcg/kg administered after each dialysis session (3 times/week)
  CR845 0.5 mcg/kg: IV medication delivered three times/week
- Double-blind Placebo: IV Placebo administered after each dialysis session (3 times/week)
  Placebo: IV medication delivered three times/week
Period: Period 1: Double-blind Phase
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo | Open-label CR845 0.5 mcg/kg
Started | 189 | 189 | 0
Completed | 162 | 170 | 0
Not Completed | 27 | 19 | 0
Period: Period 2: Open-label Phase
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo | Open-label CR845 0.5 mcg/kg
Started | 0 | 0 | 313
Completed | 0 | 0 | 189
Not Completed | 0 | 0 | 124

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo | Total
Number analyzed (Participants) | 189 | 189 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (11.16) | 56.7 (13.89) | 57.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 70 | 147
  Male | 112 | 119 | 231
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 5 | 11
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
  Black or African American | 82 | 76 | 158
  White | 91 | 93 | 184
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Itch Intensity as Assessed by the Percentage of Patients Achieving an Improvement From Baseline ≥3 Points With Respect to the Weekly Mean of the Daily 24-hour Worst Itching Intensity Numerical Rating Scale (NRS) Score at Week 12
Description: Intensity of itch will be measured using an NRS used to indicate the intensity of the worst itching over the past 24 hours using a 0 to 10 numeric rating scale, where "0" represents "no itching" and "10" represents "worst itching imaginable". LS means estimated percent, odds ratio and P value used a logistic regression model.
Time Frame: Week 12
Population: Data include one patient who had been randomly assigned to the placebo group and who withdrew from the trial before receiving the first dose of placebo.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | CR845 0.5mcg/kg | Placebo
Number analyzed (Participants) | 189 | 189
percentage of subjects | 51.0 [42.9 to 58.9] | 27.6 [20.2 to 36.6]
Statistical Analysis 1: Comparison: CR845 0.5mcg/kg vs Placebo; Test type: Superiority; p < 0.001, Cui, Hung, Wang; Odds Ratio (OR) = 2.72, 95% CI 2-sided [1.72 to 4.30]

2. Secondary Outcome: Improvement in Itch-related Quality of Life as Assessed by the Change From Baseline in 5-D Itch Scale Score at the End of Week 12
Description: The 5-D Itch Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past 2 weeks. The questions cover five dimensions of itch including the degree, duration of itch/day, direction (improvement/worsening), disability (impact on activities such as work), and body distribution of itch. The 5-D Itch Scale has 5 questions; the total 5-D Itch Scale score ranges from 5 to 25, with higher scores indicating worse responses.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo
Number analyzed (Participants) | 189 | 189
score on a scale | -5.0 [-5.7 to -4.4] | -3.7 [-4.4 to -3.1]
Statistical Analysis 1: Comparison: Double-blind CR845 0.5mcg/kg vs Double-blind Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.0 to -0.5], Standard Error of Mean 0.38

3. Secondary Outcome: Improvement in Itch-related Quality of Life as Assessed by the Change From Baseline in Total Skindex-10 Scale Score at the End of Week 12
Description: The Skindex-10 Scale is a multidimensional questionnaire which assesses itch-related quality of life over the past week. The questions cover 3 domains: disease, mood/emotional distress, and social functioning domain. The Skindex-10 has 10 questions; the total Skindex-10 score ranges from 0 to 60. A lower total score represents better quality of life.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo
Number analyzed (Participants) | 189 | 189
score on a scale | -17.2 [-19.6 to -14.7] | -12.0 [-14.5 to -9.6]
Statistical Analysis 1: Comparison: Double-blind CR845 0.5mcg/kg vs Double-blind Placebo; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-8.0 to -2.3], Standard Error of Mean 1.44

4. Secondary Outcome: Reduction of Itch Intensity as Assessed by the Percentage of Patients Achieving an Improvement From Baseline ≥4 Points With Respect to the Weekly Mean of the Daily 24-hour Worst Itching Intensity NRS Score at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo
Number analyzed (Participants) | 189 | 189
percentage of subjects | 38.9 [29.8 to 48.7] | 18.0 [12.1 to 26.0]
Statistical Analysis 1: Comparison: Double-blind CR845 0.5mcg/kg vs Double-blind Placebo; Test type: Superiority; p < 0.001, Cui, Hung, Wang; Odds Ratio (OR) = 2.89, 95% CI 2-sided [1.75 to 4.76]

ADVERSE EVENTS:
Time Frame: The period of adverse event reporting will start after the signing of the informed consent form (ICF) through the study Follow-up Visit or Early Termination Visit (or 7 days after the last dose if no Early Termination Visit was conducted).
Description: The study includes a Double-blind Phase, an Open-label Extension Phase, and a Follow-up Period. Patients who received at least 30 doses of study drug (either active or placebo) during the 12-week Double-blind Treatment Period and continue to meet other eligibility criteria will be eligible to receive open-label CR845 for an additional 52 weeks. Data exclude one patient randomized to placebo and who withdrew from the trial before receiving the first dose of placebo; no safety data collected.
Arm/Group | Double-blind CR845 0.5mcg/kg | Double-blind Placebo | Open-label CR845 0.5 mcg/kg
All-Cause Mortality (participants affected / at risk) | 2/189 | 2/188 | 22/313
Serious Adverse Events (participants affected / at risk) | 49/189 | 41/188 | 167/313
Other Adverse Events (participants affected / at risk) | 40/189 | 30/188 | 205/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind CR845 0.5mcg/kg (N=189) | Double-blind Placebo (N=188) | Open-label CR845 0.5 mcg/kg (N=313)
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 3
Angina pectoris (Cardiac disorders) | 2 | 0 | 5
Bradycardia (Cardiac disorders) | 0 | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 11
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 5
Angina unstable (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 6
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 6
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3
Chest pain (General disorders) | 1 | 3 | 3
Asthenia (General disorders) | 2 | 0 | 8
Complication associated with device (General disorders) | 1 | 0 | 8
Gait inability (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 5 | 23
Sepsis (Infections and infestations) | 3 | 4 | 10
Septic shock (Infections and infestations) | 1 | 3 | 6
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 6
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 1
Enterobacter bacteraemia (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 4
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 4
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 3
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 2
Complications of transplanted liver (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 5
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 6
Troponin increased (Investigations) | 0 | 2 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 4 | 12
Fluid overload (Metabolism and nutrition disorders) | 2 | 4 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 2 | 10
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 2
Seizure (Nervous system disorders) | 1 | 1 | 4
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 2 | 9
Delusional disorder, unspecified type (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 1 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 10
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 3 | 2 | 8
Aneurysm arteriovenous (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 8
Thrombosis (Vascular disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 2
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 0 | 1
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 3
Ascities (Gastrointestinal disorders) | 0 | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 7
Death (General disorders) | 0 | 0 | 3
Hernia (General disorders) | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 3
Influenza (Infections and infestations) | 0 | 0 | 3
Cystitis (Infections and infestations) | 0 | 0 | 2
Device related infection (Infections and infestations) | 0 | 0 | 2
Osteomyelitis acute (Infections and infestations) | 0 | 0 | 2
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 2
Anal abscess (Infections and infestations) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1
Mastitis (Infections and infestations) | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1
Perineal cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 1
Pyelitis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 3
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 2
Anticoagulation drug level below therapeutic (Investigations) | 0 | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1
Cacliphylaxis (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chronic kidney disease-mineral and bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 8
Encephalopathy (Nervous system disorders) | 0 | 0 | 4
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Thoracic outlet syndrome (Nervous system disorders) | 0 | 0 | 1
Uraemic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Device occlusion (Product Issues) | 0 | 0 | 1
Stent malfunction (Product Issues) | 0 | 0 | 1
Confabulation (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 0 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 11
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Loss of personal independence in daily activities (Social circumstances) | 0 | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0 | 2
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Dry gangrene (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Venous occlusion (Vascular disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind CR845 0.5mcg/kg (N=189) | Double-blind Placebo (N=188) | Open-label CR845 0.5 mcg/kg (N=313)
Diarrhoea (Gastrointestinal disorders) | 18 | 10 | 61
Nasopharyngitis (Infections and infestations) | 6 | 14 | 31
Dizziness (Nervous system disorders) | 13 | 3 | 35
Vomiting (Gastrointestinal disorders) | 10 | 6 | 43
Nausea (Gastrointestinal disorders) | 7 | 9 | 54
Fall (Injury, poisoning and procedural complications) | 6 | 8 | 50
Hypotension (Vascular disorders) | 7 | 4 | 49
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 36
Headache (Nervous system disorders) | 8 | 4 | 36
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 3 | 35
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 8 | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 34
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5 | 31
Constipation (Gastrointestinal disorders) | 6 | 4 | 29
Hypertension (Vascular disorders) | 7 | 6 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 25
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 23
Upper respiratory tract infection (Infections and infestations) | 7 | 1 | 20
Pyrexia (General disorders) | 5 | 2 | 17
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 16
Anxiety (Psychiatric disorders) | 3 | 2 | 16
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03422653/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03422653/SAP_001.pdf